CLINICAL TRIAL: NCT07331675
Title: Effects of Marble Play on Hand Grip Strength and Handwriting Skills Among School Going Children
Brief Title: Effect of Marble Play on Handgrip Strength and Handwriting Among School Going Children.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: maqsood Bibi
Record Dates: First submitted 2025-12-29; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Hand Grasp
Keywords: Dynamometer; Hand writing skills; Hand grip strength

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Marble play group (Experimental): The experimental group will participate in one-on-one sessions of Marble Play game with progressive difficulty levels, designed to enhance fine motor control, handgrip and handwriting skills.
  Interventions: Other: Marble play game
- Free play (Other): The control group will continue with their regular free play activities.
  Interventions: Other: Free Play

INTERVENTIONS:
Other: Marble play game — Participants have to be sure to play in playground, as we will used natural ground floor. A small circle will be dig. A straight line will be marked 40 cm away from the edge of the circle. At the beginning of game, the researcher will place 10 target marbles in the circle. The participant will be given a marble.
  Arms: Marble play group
Other: Free Play — The control group (n=38) will continues regular playing activities except Marble play.
  Arms: Free play

SUMMARY:
This study aims to address the effects of a Marble Play on the handgrip strength and handwriting skills of primary school children, providing empirical evidence for a cost-effective and culturally relevant therapeutic tool. This study will be a randomized controlled trial. A total of 46 children from Grades 1-3 will be recruited via convenience sampling and randomly assigned to either an experimental group (n=23) or a control group (n=23).The experimental group will participate in one-on-one sessions of Marble Play game with

.The control group will continue with their regular free play activities. The primary assessment tools will be the Evaluation Tool of Children's Handwriting (ETCH) to measure writing legibility and speed, and a hand-held dynamometer to measure hand grip strength.

DETAILED DESCRIPTION:
In 2022, Audrey Saile and Mohd Hanafi Mohd Yasin hey conducted a study in Malaysia, to investigate the efficacy of fine motor training for improving handwriting legibility among students with special educational needs. Their study used a quasi-experimental pre-test/post test design but was limited by a very small, purposefully selected sample of only four students.

Despite this limitation, the results indicated a positive outcome: the treatment group showed an average 15-point increase on a modified Handwriting Legibility Scale, improving their performance from "very poor" to "moderate." The authors concluded that fine motor training is a valuable intervention for enhancing the handwriting skills of SEN students.

Current literature reveals a significant gap in research examining marble play as a targeted fine motor intervention. While existing studies have explored the effectiveness of various manipulative activities such as clay modeling, bead threading, and drawing exercises for fine motor development, there is a notable absence of research that specifically isolates and examines the unique benefits of marble play. This represents a critical oversight, given the accessibility and affordability of marbles as intervention tool. The findings of this study will provide much-needed, evidence-based guidance for educators and therapists, particularly those working in resource-limited environments.

ELIGIBILITY:
Inclusion Criteria:

* Children enrolled in Grade 1-3 (typically aged 6-9 years)
* Children with normal cognitive development, as assessed by school records or teacher reports
* Students with average or below average handwriting fluency (based on teacher observation or pre-test).
* Parental or guardian consent obtained for participation.
* Regular school attendance and ability to participate in intervention sessions.

Exclusion Criteria:

* Children with significant visual or motor impairments that may affect fine motor coordination.
* Participants with a known history of dust allergy or diagnosed allergic rhinitis triggered by dust exposure will be excluded.
* Individuals with a current or recent (within the last 6 months) fracture of any upper, wrist, or hand) will be excluded.
* Students with a history of behavioral issues that would prevent consistent participation in structured play.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 46 (Estimated)
Dates: Start 2025-12-22 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
Hand Grip Strength | Baseline and after 6 weeks
  Hand grip strength will be measured by dynamometer
handwriting skills | Baseline and after 6 weeks
  handwriting skills will be measured by ECTH. ECTH scoring refers to the Evaluation Tool of Children's Handwriting (ECTH), a criterion-referenced assessment for grades 1-6, scored by occupational therapists and educators to evaluate manuscript/cursive writing speed and legibility (letter/word formation, size, spacing, alignment) through specific tasks like copying, dictation, and sentence composition, yielding scores for each task and overall legibility percentages, with established cutoffs (e.g., Total Letter <90%, Total Word <85%) indicating dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Aamna Hassan, MS, Principal Investigator — Riphah International University, Lahore
Locations (1):
- Aamna Hassan, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hendrickx S. The adolescent and adult neuro-diversity handbook: Asperger's syndrome, ADHD, dyslexia, dyspraxia, and related conditions: Jessica Kingsley Publishers; 2010.
- [Background] Davis RD, Braun EM. The Gift of Learning: Proven New Methods for Correcting ADD, Math & Handwriting Problems: Penguin; 2003.
- [Background] Engel-Yeger B, Nagauker-Yanuv L, Rosenblum S. Handwriting performance, self-reports, and perceived self-efficacy among children with dysgraphia. Am J Occup Ther. 2009 Mar-Apr;63(2):182-92. doi: 10.5014/ajot.63.2.182. PMID 19432056